CLINICAL TRIAL: NCT05821556
Title: Randomized Phase 2 Study of Valproic Acid combinEd With Simvastatin and Gemcitabine/Nab-paclitaxel-based Regimens in Untreated Metastatic Pancreatic Adenocarcinoma Patients (The VESPA Trial).
Brief Title: Valproic Acid/Simvastatin Plus Gemcitabine/Nab-paclitaxel Based Regimens in Untreated Metastatic Pancreatic Adenocarcinoma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VESPA; 1/23 (Other: IRCCS I.N.T. "G. Pascale")
Record Dates: First submitted 2023-03-23; First posted 2023-04-20 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Adenocarcinoma of the Pancreas
Keywords: Metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Valproic Acid; Simvastatin; Gemcitabine; Taxes; Cisplatin; Capecitabine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized electronically 1:1 to one of the two arms:
  A. Standard: Nab-paclitaxel 125 mg/m2 followed by gemcitabine 1000 mg/m2 on days 1, 8, and 15 (AG); or nab-paclitaxel 150 mg/m2, followed by gemcitabine 800 mg/m2, followed by cisplatin 30 mg/m2 on days 1 and 15, and oral capecitabine 1250 mg/m2 on days 1-28 (PAXG). B. Experimental: Chemotherapy (AG or PAXG) + simvastatin oral daily at a fixed dosage of 20 mg in combination with increasing doses of valproic acid administered oral daily from day -7 with an intra-patient titration for a final target serum level of 50-100µg/ml.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard (Active Comparator): Nab-paclitaxel 125 mg/m2 followed by gemcitabine 1000 mg/m2 on days 1, 8, and 15 (AG); or nab-paclitaxel 150 mg/m2, followed by gemcitabine 800 mg/m2, followed by cisplatin 30 mg/m2 on days 1 and 15, and oral capecitabine 1250 mg/m2 on days 1-28 (PAXG).
  Interventions: Drug: Gemcitabine 1000 mg; Drug: Nab paclitaxel; Drug: Cisplatin; Drug: Capecitabine
- Experimental (Experimental): Chemotherapy (AG or PAXG) + simvastatin oral daily at a fixed dosage of 20 mg in combination with increasing doses of valproic acid administered oral daily from day -7 with an intra-patient titration for a final target serum level of 50-100µg/ml.
  Interventions: Drug: Valproic acid; Drug: Simvastatin 20mg; Drug: Gemcitabine 1000 mg; Drug: Nab paclitaxel; Drug: Cisplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Valproic acid — The treatment should be started within 3 days from randomization. One cycle consisted of 28 days of treatment for both arms. Patients will continue to receive study treatment up to 6 cycles until disease progression, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria. Continuation of treatment, over the six cycles, will be allowed only in case of clinical benefit, defined as continuous decrease of CA19-9 concentration or radiological response, without unacceptable toxicity.
  All subjects who finish treatment, whichever the reason, will enter in the follow-up. We expect that for the primary endpoint, PFS, follow-up will last up to 10 months after enrollment.
  Anyhow, all subjects will be followed until death and data on subsequent treatment will be collected.
  Arms: Experimental
Drug: Simvastatin 20mg — The treatment should be started within 3 days from randomization. One cycle consisted of 28 days of treatment for both arms. Patients will continue to receive study treatment up to 6 cycles until disease progression, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria. Continuation of treatment, over the six cycles, will be allowed only in case of clinical benefit, defined as continuous decrease of CA19-9 concentration or radiological response, without unacceptable toxicity.
  All subjects who finish treatment, whichever the reason, will enter in the follow-up. We expect that for the primary endpoint, PFS, follow-up will last up to 10 months after enrollment.
  Anyhow, all subjects will be followed until death and data on subsequent treatment will be collected.
  Arms: Experimental
Drug: Gemcitabine 1000 mg — The treatment should be started within 3 days from randomization. One cycle consisted of 28 days of treatment for both arms. Patients will continue to receive study treatment up to 6 cycles until disease progression, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria. Continuation of treatment, over the six cycles, will be allowed only in case of clinical benefit, defined as continuous decrease of CA19-9 concentration or radiological response, without unacceptable toxicity.
  All subjects who finish treatment, whichever the reason, will enter in the follow-up. We expect that for the primary endpoint, PFS, follow-up will last up to 10 months after enrollment.
  Anyhow, all subjects will be followed until death and data on subsequent treatment will be collected.
Drug: Nab paclitaxel — The treatment should be started within 3 days from randomization. One cycle consisted of 28 days of treatment for both arms. Patients will continue to receive study treatment up to 6 cycles until disease progression, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria. Continuation of treatment, over the six cycles, will be allowed only in case of clinical benefit, defined as continuous decrease of CA19-9 concentration or radiological response, without unacceptable toxicity.
  All subjects who finish treatment, whichever the reason, will enter in the follow-up. We expect that for the primary endpoint, PFS, follow-up will last up to 10 months after enrollment.
  Anyhow, all subjects will be followed until death and data on subsequent treatment will be collected.
Drug: Cisplatin — The treatment should be started within 3 days from randomization. One cycle consisted of 28 days of treatment for both arms. Patients will continue to receive study treatment up to 6 cycles until disease progression, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria. Continuation of treatment, over the six cycles, will be allowed only in case of clinical benefit, defined as continuous decrease of CA19-9 concentration or radiological response, without unacceptable toxicity.
  All subjects who finish treatment, whichever the reason, will enter in the follow-up. We expect that for the primary endpoint, PFS, follow-up will last up to 10 months after enrollment.
  Anyhow, all subjects will be followed until death and data on subsequent treatment will be collected.
Drug: Capecitabine — The treatment should be started within 3 days from randomization. One cycle consisted of 28 days of treatment for both arms. Patients will continue to receive study treatment up to 6 cycles until disease progression, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria. Continuation of treatment, over the six cycles, will be allowed only in case of clinical benefit, defined as continuous decrease of CA19-9 concentration or radiological response, without unacceptable toxicity.
  All subjects who finish treatment, whichever the reason, will enter in the follow-up. We expect that for the primary endpoint, PFS, follow-up will last up to 10 months after enrollment.
  Anyhow, all subjects will be followed until death and data on subsequent treatment will be collected.

SUMMARY:
This is a proof-of-concept, Open label, randomized, multicentric, superiority phase-2 study.

DETAILED DESCRIPTION:
The study hypothesizes that valproic acid (VPA) in combination with simvastatin (SIM) may improve the efficacy of first-line gemcitabine and nab-paclitaxel-based regimens and extend progression free survival (PFS) as compared with chemotherapy alone, in patients with metastatic pancreatic ductal adenocarcinoma (mPDAC).

Correlative studies on tumor and blood samples could identify potential biomarkers of toxicity and efficacy helping to define personalized treatment strategy and adding new insight into the antitumor mechanism of the combination approach.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to study procedures and to correlative studies.
2. Histologically or cytologically proven metastatic PDAC.
3. No prior treatments (chemotherapy, radiation or surgery) for PDAC
4. Either sex aged ≥ 18 years.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1 at study entry.
6. Imaging-documented measurable disease, according to RECIST 1.1 criteria.
7. Known dihydropyrimidine dehydrogenase (DPD) activity is mandatory for patients enrolled in PAXG scheme.
8. Adequate bone marrow haematological function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L AND platelet count ≥ 100 x 109/L AND haemoglobin ≥ 9 g/dL.
9. Adequate liver function: total bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 2 in case of biliary stent) and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 5 X ULN.
10. Adequate renal function: serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min in males and ≥50 mL/min in females (calculated according to Cockroft-Gault formula).

Exclusion Criteria:

1. Prior malignancy within one year. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
2. Prior chemotherapy or any other medical treatment for metastatic PDAC (previous adjuvant chemotherapy is allowed if terminated > 6 months previously).
3. Patients who have had prior treatment with an HDAC inhibitor and patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid.
4. Current use of statins or fibrates or any medication for hypercholesterolemia for any time during the 3 months before the study.
5. Proven hypersensitivity to statins and to any component of the other medications used in the trial.
6. Major surgical intervention within 4 weeks prior to enrollment;
7. Pregnancy and breast-feeding.
8. Brain metastasis.
9. Hepatitis or any severe liver disorder.
10. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study, or which would jeopardize compliance with the protocol, or would interfere with the results of the study.
11. Patients with long QT-syndrome or QTc interval duration > 480 msec or concomitant medication with drugs prolonging QTc (see list in the appendix).
12. History of poor co-operation, non-compliance with medical treatment, unreliability or any condition that may impair the patient's understanding of the Informed consent form.
13. Participation in any interventional drug or medical device study within 30 days prior to treatment start.
14. Patients who cannot take oral medication, who require intravenous alimentation, have had prior surgical procedures affecting absorption, or have active peptic ulcer disease.
15. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study and until 6 months after the last trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 40 months
  PFS is defined as the time from randomization to the first documentation of objective disease progression by RECIST 1.1 criteria, or death due to any cause, whichever occurs first. PFS will be censored at the time of the last available tumor assessment documenting absence of progressive disease for patients alive at the time of analysis.

SECONDARY OUTCOMES:
Objective Tumor Response Rate (ORR) | 40 months
  Objective Tumor Response Rate (ORR) as defined by RECIST 1.1, calculated as the proportion of patients achieving complete or partial response relative to total enrolled patients.
Duration of Objective response (DOR) | 40 months
  Duration of Objective response (DOR) defined as the first occurrence of a documented objective response until progression or death for any cause.
Disease Control Rate (DCR) | 40 months
  Disease Control Rate (DCR) defined as the proportion of patients with complete/partial response and stable disease as their best response.
Overall Survival (OS) | 40 months
  Overall Survival (OS) defined as the time from randomization to the date of death due to any cause. OS will be censored at the last date the patient was known to be alive for patients alive at the time of analysis.
Overall toxicity rate | 40 months
  Overall toxicity rate defined as the proportion of patients experiencing any grade AE accordingly to the NCI Common Terminology Criteria of Adverse Events (NCI CTC-AE) Version 5, relative to the total of patients receiving at least one cycle of treatment.AE will be listed individually by the patient and summarized overall (severity grades 1-4) and for grade ≥3 by treatment received.
Quality of Life (QoL) | 40 months
  Quality of Life (QoL), based on questionnaire EORTC QLQ-C30 at baseline (prior to treatment start, once eligibility is confirmed) and every 8 weeks until 40 weeks after randomization, regardless of disease progression, or death

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Budillon, Principal Investigator — IRCCS I.N.T. "G. Pascale; Antonio Avallone, Principal Investigator — IRCCS I.N.T. "G. Pascale
Locations (5):
- Italy (4):
  - Istituto Nazionale Tumori di Napoli - IRCCS - Fondazione G. Pascale, Napoli, Italy
  - Università vita e Salute, IRCCS San Raffaele, Milan, Milano
  - Università Cattolica Del Sacro Cuore, IRCCS Fondazione Policlinico Universitario Gemelli - Medical Oncology, Roma, Italia, Roma, Roma
  - University of Verona Hospital Trust, Verona, Verona
- Ramon y Cajal Hospital and Health Research Institute (IRYCIS), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Budillon A, Leone A, Passaro E, Silvestro L, Foschini F, Iannelli F, Roca MS, Macchini M, Bruzzese F, Garcia Bermejo ML, Rodriguez Garrote M, Tortora G, Milella M, Reni M, Fuchs C, Hewitt E, Kubiak C, Di Gennaro E, Giannarelli D, Avallone A. Randomized phase 2 study of valproic acid combined with simvastatin and gemcitabine/nab-paclitaxel-based regimens in untreated metastatic pancreatic adenocarcinoma patients: the VESPA trial study protocol. BMC Cancer. 2024 Sep 19;24(1):1167. doi: 10.1186/s12885-024-12936-w. PMID 39300376